CLINICAL TRIAL: NCT03145246
Title: Long-Term Outcome Following Regenerative Periodontal Treatment of Intrabony Defects: A Retrospective Study at Mahidol University
Brief Title: Long-Term Outcome Following Regenerative Periodontal Treatment of Intrabony Defects
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/DT105
Record Dates: First submitted 2015-11-13; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Regenerative Periodontal Treatment
Keywords: intrabony defect; periodontal regeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- tooth loss: regeneration treated teeth loss
  Interventions: Procedure: regeneration treated teeth loss
- clinical attachment loss ≥ 2 mm: regenerated treated teeth with clinical attachment loss ≥ 2 mm
  Interventions: Procedure: regenerated treated teeth with clinical attachment loss
- clinical attachment loss loss < 2 mm: regenerated treated teeth with clinical attachment loss < 2 mm
  Interventions: Procedure: regenerated treated teeth with clinical attachment loss

INTERVENTIONS:
Procedure: regeneration treated teeth loss — number of regeneration treated teeth loss
  Groups: tooth loss
Procedure: regenerated treated teeth with clinical attachment loss — regenerated treated teeth with clinical attachment loss ≥ 2 mm
  Groups: clinical attachment loss loss < 2 mm; clinical attachment loss ≥ 2 mm

SUMMARY:
Many years ago, periodontal regenerative treatment has been done in Periodontics and Oral Medicine Clinic, Faculty of Dentistry, Mahidol University, Bangkok, Thailand. However, there is still lacking of study about long-term result of periodontal regenerative treatment of intrabony defects.

DETAILED DESCRIPTION:
Beside, in the present, some materials for periodontal regenerative treatment are still expensive. Periodontists and patients have to plan together based on not only rationale of treatment but also cost and effectiveness. Thus the long-term result of treatment could be useful for the decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received regenerative therapy of the intrabony defects
* Patients who had the record of re-evaluation at 1 year post-surgery

Exclusion Criteria:

* Patients who received regenerative therapy involving the furcation area
* Patients who received non-periodontal regenerative therapy
* Patients who received endodontic regeneration
* Patients who had an incomplete periodontal data recording

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients who received regenerative periodontal therapy of the intrabony defects by post-graduate students at the Periodontics and Oral Medicine Clinic, Faculty of Dentistry, Mahidol University, Thailand and were placed in the Recall Patient Bank from 2000 to 2014.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of regenerative-treated tooth loss after periodontal regeneration | 1 year
  Percentage of regenerative-treated tooth loss since 1 year after periodontal regeneration until last visit of supportive periodontal treatment
Percentage of regenerative-treated sites with clinical attachment loss ≥ 2 mm | 1 year
  Percentage of regenerative-treated sites with clinical attachment loss ≥ 2 mm since 1 year after periodontal regeneration until last visit of supportive periodontal treatment

SECONDARY OUTCOMES:
Variables (patient and tooth characteristics) that associated with tooth loss or clinical attachment loss | 1 year
  Patient variables and tooth characteristics associated with regenerative-treated tooth loss or sites with clinical attachment loss ≥ 2 mm from any supportive periodontal treatment visits (the last supportive periodontal treatment visit) compared to baseline or 1-year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kanyawat Rattanasuwan, Study Director — Mahidol University

IPD SHARING:
Plan to Share IPD: No